CLINICAL TRIAL: NCT00128180
Title: A Phase II Randomized, Double-Blind, Placebo-Controlled Trial of Intravenous Methylprednisolone as a Treatment for Presumed Hantavirus Cardiopulmonary Syndrome
Brief Title: Efficacy of Methylprednisolone for Hantavirus Cardiopulmonary Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-010; U19 A1045452
Record Dates: First submitted 2005-08-05; First posted 2005-08-09 (Estimated); Results first posted 2012-07-10 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Hantavirus Infections
Keywords: hantaviruses, methylprednisolone, cardiopulmonary syndrome
MeSH Terms: conditions — Hantavirus Infections; Hantavirus Pulmonary Syndrome | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Active Comparator): Methylprednisolone
  Interventions: Drug: Methylprednisolone
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylprednisolone — Intravenous methylprednisolone 16 mg/kg/day for 3 days as follows: 8 mg/kg (up to 500 mg) given over first hour followed by 8 mg/kg over the next 23 hours; then 16 mg/kg (up to 1000 mg) on days 2 and 3 administered over 24 hours.
  Other Names: Medrol
  Arms: Active
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if a drug, called methylprednisolone, is safe and effective in people with Hantavirus infection. Individuals 2 years of age or older are invited to participate in this study if their doctor suspects or knows they have Hantavirus infection. Volunteers will either be given methylprednisolone or placebo (contains no medication) through a needle inserted in a vein for 3 days. During the first 7 days of hospitalization procedures may include blood tests, physical exams, chest x-rays, and urine tests. During study visits on days 14, 28, 84 and 180 after diagnosis, the doctors will ask about health, examine the body, take a chest X-ray, collect blood for safety testing and for measuring antibodies, and do breathing tests on volunteers. Participants will be involved in the study for about 6 months.

DETAILED DESCRIPTION:
This study is a phase II, randomized, double-blind, placebo-controlled evaluation of intravenous methylprednisolone versus placebo in treatment of hantavirus cardiopulmonary syndrome (HCPS). Patients with suspected or known hantavirus will be randomized to receive intravenous methylprednisolone or placebo over 3 days. Following the completion of this acute phase therapy, patients will be seen for follow up visits on days 14, 28, 84 and 6 months after study entry. Follow up visits will include a physical examination, including vital signs. In addition, blood will be drawn for a blood count, clinical chemistries, and quantitative polymerase chain reaction (day 14). Since Hantavirus pathogenesis involves the pulmonary system, other tests to be performed include chest x ray (day 28) and spirometry (days 28 and 180). The study will require 60 subjects with confirmed Hantavirus infection. Study subjects will include males and females greater than or equal to 2 years of age suspected of having Hantavirus disease. The enrolling co investigator must feel that Hantavirus disease is likely on the basis of the clinical syndrome. The primary study objectives are to: assess the efficacy of intravenous methylprednisolone in reducing the severity of HCPS and assess the safety of methylprednisolone in persons with suspected and proven Hantavirus infection. The secondary objectives are to: assess the impact of therapy on viremia and assess whether measurement of neutralizing antibody titers at entry or Human Leukocyte Antigen (HLA) typing can identify subgroups with increased risk of severe disease and/or death and whether therapy is effective in these subgroups. The primary endpoints will include: the proportion of subjects who develop one or more of the following critical events associated with severe disease 28 days after study entry: death, PaO2/FiO2 ratio less than or equal to 55, cardiac index less than or equal to 2.2, pulseless electrical activity, ventricular tachycardia or fibrillation; and number of serious adverse events determined by study investigators to be at least possibly related to study treatment. For this endpoint researchers will report: the median number of serious adverse events and the proportion that experience one or more serious adverse events. The secondary study endpoints include: to assist in defining the natural history of the disease but will not meaningfully affect treatment: Extracorporeal Membrane Oxygenation (ECMO); duration of intensive care unit stays; duration of hospital stays; duration of shock and/or pressor/inotropic support; length of time on mechanical ventilation; intubated and placed on a ventilator; refractory shock despite fluid resuscitation; and serum creatinine greater than or equal to 3.0 milligrams/deciliter.

ELIGIBILITY:
Inclusion Criteria:

Informed consent is given by patient or guardian.

And one of the following:

* Confirmed diagnosis: Positive hantavirus IgM assay or detection of hantavirus in plasma or serum by RT-PCR in the presence of an acute febrile illness of less than 12 days duration, and

  1. Onset of hypoxia (oxygen saturation less than or equal to 92% or requiring supplemental oxygen) one or more days after onset of symptoms, and
  2. Development of pulmonary infiltrates on chest X-ray. OR
* Presumptive diagnosis: The presumptive diagnosis of acute hantavirus disease of less than 12 days duration with:

  1. Febrile illness (subjective or documented) in the judgment of the enrolling investigator; and
  2. Headache or myalgia or at least one digestive symptom (nausea, diarrhea, vomiting, abdominal pain) and
  3. A platelet count less than 150,000 on peripheral smear; and
  4. Onset of hypoxia (oxygen saturation less than or equal to 92% or requiring supplemental oxygen) one or more days after onset of symptoms, and
  5. Development of bilateral pulmonary infiltrates on chest X-ray

Exclusion Criteria:

* Age less than 2 years.
* If presumptive diagnosis is the inclusion criteria: subjects with a likely diagnosis other than hantavirus infection, including any positive culture or direct test for respiratory viruses (e.g., influenza, RSV, etc) or group A Streptococcus in a person with an illness compatible with streptococcal pharyngitis, a positive culture from a normally sterile site, or a presentation consistent with bacterial pneumonia.
* Immunocompromised patients at risk of opportunistic infection (e.g., patients with HIV infection, underlying malignancy, or who have received chemotherapy or immunosuppressive drugs within 30 days.)
* Patients who have or will receive any systemic antiviral medication (other than acyclovir, famciclovir, amantadine or rimantadine), systemic corticosteroids equivalent to approximately 0.5mg/kg prednisone, or any investigational drug within 30 days before enrollment or during treatment.
* Any period of extreme bradycardia, pulseless electric activity
* Active GI bleeding, with hematemesis, melena or hematochezia or documented by upper or lower endoscopy or by gastric aspiration.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2003-01; Primary Completion 2010-12 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Vial, MD, Principal Investigator — Universidad del Desarrollo
Locations (1):
- Facultad de Medicina Clinica Alemana- Universidad del Desarrollo, Santiago, Chile

REFERENCES:
- [Result] Vial PA, Valdivieso F, Ferres M, Riquelme R, Rioseco ML, Calvo M, Castillo C, Diaz R, Scholz L, Cuiza A, Belmar E, Hernandez C, Martinez J, Lee SJ, Mertz GJ; Hantavirus Study Group in Chile. High-dose intravenous methylprednisolone for hantavirus cardiopulmonary syndrome in Chile: a double-blind, randomized controlled clinical trial. Clin Infect Dis. 2013 Oct;57(7):943-51. doi: 10.1093/cid/cit394. Epub 2013 Jun 19. PMID 23784924

RESULTS

PARTICIPANT FLOW:
Groups:
- Active: Active drug
- Placebo: Placebo group
Period: Overall Study
Arm/Group | Active | Placebo
Started | 32 | 34
Completed | 32 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 32 | 34 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 6 | 9
  Between 18 and 65 years | 28 | 27 | 55
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.94 (15.49) | 36.26 (15.13) | 38.53 (15.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 22 | 24 | 46
Region of Enrollment [Number; unit: participants]
  Chile | 32 | 34 | 66

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Who Develop Death, PaO2/FiO2 Ratio Less Than or Equal to 55, Cardiac Index Less Than or Equal to 2.2, Pulseless Electrical Activity, Ventricular Tachycardia or Fibrillation
Time Frame: 28 days
Population: Per protocol, the efficacy analysis was limited to participants with confirmed hantavirus infection.
Measure: Number; unit: proportion of paticipants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 30 | 30
proportion of paticipants | 0.27 [0.12 to 0.46] | 0.47 [0.28 to 0.65]
Statistical Analysis 1: Comparison: Active vs Placebo; Test type: Superiority or Other; p = 0.18, Fisher Exact

2. Primary Outcome: Number of Participants With SAEs
Description: The Number of participants with SAEs
Time Frame: 6 months
Population: Per protocol, safety analysis inluded all participants, including those where hantavirus infection was not confirmed.
Measure: Number; unit: participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 32 | 34
participants | 14 | 25

3. Secondary Outcome: Number of Participants on Extracorporeal Membrane Oxygenation (ECMO)
Description: number of participants
Time Frame: 6 months
Population: Per protocol, efficacy analysis was limited to participants with confirmed hantavirus infection.
Measure: Number; unit: participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 30 | 30
participants | 0 | 0

4. Secondary Outcome: Duration of ICU Stays
Time Frame: 6 months
Population: Per protocol, efficacy analysis was limited to participants with confirmed hantavirus infection, and this analysis was limited to those who were admitted to ICU. Four subjects with confirmed hantavirus infection were not admitted to ICU.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Active | Placebo
Number analyzed (Participants) | 27 | 29
days | 4.48 (2.78) | 5.83 (4.43)

5. Secondary Outcome: Duration of Hospital Stay in Days
Description: Days
Time Frame: 6 months
Population: Per protocol, efficacy analysis was limited to participants with confirmed hantairus infection.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Active | Placebo
Number analyzed (Participants) | 30 | 30
days | 8.90 (6.08) | 10.67 (8.93)

6. Secondary Outcome: Duration of Shock and/or Pressor/Inotropic Support
Description: Pressor/inotropic support refers to the use of adrenaline-like medications to maintain blood pressure and cardiac output.
Time Frame: 6 months
Population: Per protocol, efficacy analysis was limited to participants with confirmed hantavirus infection.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Active | Placebo
Number analyzed (Participants) | 30 | 30
days | 2.67 (2.10) | 3.75 (3.23)

7. Secondary Outcome: Number of Participants Intubated and Placed on a Ventilator After Study Entry.
Description: Participants
Time Frame: 6 months
Population: This efficacy this analysis was limited to participants with confirmed hantavirus infection who were not already intubated at study entry.
Measure: Number; unit: participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 26 | 20
participants | 6 | 10

8. Secondary Outcome: Number of Participants Who Developed Refractory Shock Despite Fluid Resuscitation After Study Entry
Description: Refractory shock refers to shock that persists despite fluid resucitation. Fluid resusitation refers to administration of intravenous fluids to maintain blood pressure and cardiac output.
Time Frame: 6 months
Population: Per protocol, this efficacy analysis was limited to participants with confirmed hantavirus infection who were not already in shock at study entry.
Measure: Number; unit: participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 21 | 15
participants | 4 | 6

9. Secondary Outcome: Length of Time on a Ventilator
Time Frame: 6 months
Population: Per protocol this efficacy analysis was limited to participants with confirmed hantavirus infection who were intubated and on a ventillator.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Active | Placebo
Number analyzed (Participants) | 11 | 20
days | 2.64 (2.06) | 4.95 (4.48)

10. Secondary Outcome: Development of Serum Creatinine Greater Than or Equal to 3.0 mg/dL After Study Entry
Time Frame: 6 months
Population: Per protocol, this efficay analysis was limited to participants with confirmed hantavirus infection who did not have a serum creatinine equal or greater to 3.0 mg/dL at entry.
Measure: Number; unit: participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 29 | 30
participants | 1 | 6

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Active | Placebo
Serious Adverse Events (participants affected / at risk) | 14/32 | 25/34
Other Adverse Events (participants affected / at risk) | 14/32 | 20/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=32) | Placebo (N=34)
Blood and lymphatic (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cardiac disorder (Cardiac disorders) | 7 (7) | 19 (19)
Hepatobiliary disorders (Hepatobiliary disorders) | 11 (11) | 15 (15)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Nervous system disorders (Nervous system disorders) | 1 (1) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 4 (4)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=32) | Placebo (N=34)
Eye Disorder (Eye disorders) | 0 (0) | 1 (1)
Gastrointestinal Disorder (Gastrointestinal disorders) | 10 (10) | 16 (16)
General disorders (General disorders) | 3 (3) | 8 (8)
Head, Ears, Nose, Throat (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Infections and (Infections and infestations) | 0 (0) | 3 (3)
Musculoskeletal, connective tissue and bone disord (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Psychiatric Disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Vascular disorders (Vascular disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
While the study reached the target accrual of 60 confirmed cases, it was not powered to detect a difference in mortality. Higher disease severity in the placebo group at entry complicated both the efficacy and safety analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes